CLINICAL TRIAL: NCT06940739
Title: A Phase 1/2, Open-label Study of a Modified Interleukin-2 Fusion Protein (IOV-3001) in Participants With Previously Treated, Unresectable or Metastatic Melanoma Who Will Receive Lifileucel
Brief Title: A Study to Investigate the Safety and Efficacy of IOV-3001 in Adults With Advanced Melanoma Who Will Receive Lifileucel
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IOV-IL2-101
Record Dates: First submitted 2025-04-08; First posted 2025-04-23 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-05

CONDITIONS: Unresectable Melanoma; Metastatic Melanoma; Ocular Melanoma
Keywords: Tumor Infiltrating Lymphocytes; TIL; Unresectable Melanoma; Metastatic Melanoma; Cell Therapy; Autologous Adoptive Cell Therapy; Cellular Immuno-therapy; IL-2; Autologous Adoptive Cell Transfer; Melanoma; Lifileucel; Stage IV Melanoma; Malignant Melanoma; Uveal Melanoma
MeSH Terms: conditions — Melanoma; Uveal Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental): Dose escalation participants with unresectable or metastatic melanoma
  Interventions: Biological: IOV-3001

INTERVENTIONS:
Biological: IOV-3001 — IOV-3001 will be administered as a single dose by IV infusion, which will be administered in a hospital setting.

SUMMARY:
A Phase 1/2, open-label study of a modified interleukin-2 fusion protein (IOV 3001) in participants with previously treated, unresectable or metastatic melanoma who will receive lifileucel.

DETAILED DESCRIPTION:
This study is the first-in-human (FIH) study of IOV-3001. IOV-3001 is an antibody interleukin-2 (IL-2) fusion protein in which a modified form of aldesleukin is incorporated into the antibody palivizumab.

The Phase 1 portion will include 2 parts. Participants will receive IOV-3001 either before the Lifileucel regimen (Part 1) or after Lifileucel instead of aldesleukin (Part 2).

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 years of age at the time of signing the informed consent.
2. Participant has unresectable or metastatic melanoma.
3. Participant has melanoma not of uveal/ocular origin and experienced documented radiographic disease progression during systemic therapy with a PD-1/PD-L1 blocking antibody or within 12 weeks after the last dose of the PD-1/PD-L1 blocking antibody. If the tumor is BRAF V600 mutation positive, the participant also received or refused a BRAF inhibitor with or without a MEK inhibitor.

   OR Phase 1, Part 1 only: For participants with uveal melanoma, tebentafusp must have been received if available as standard of care (human leukocyte antigen [HLA]-A*02:01 positive participant and approved by local authorities for uveal melanoma) or refused.
4. Participant has an ECOG performance status of 0 or 1 and, in the investigator's opinion, an estimated life expectancy of > 6 months.
5. Phase 1, Part 2 only: Following tumor resection for lifileucel generation, the participant will have at least one remaining measurable lesion, as defined by RECIST v1.1.
6. Participant has recovered from all prior anticancer treatment-related AEs

Exclusion Criteria:

1. Participant has symptomatic untreated brain metastases.
2. Participant is at an increased risk for systemic infections; seizure disorders; coagulation disorders; or other active major medical illnesses of the cardiovascular, respiratory, or immune systems.
3. Participant has active uveitis that requires active treatment.
4. Participant has any form of primary immunodeficiency (e.g., severe combined immunodeficiency disease [SCID] or AIDS).
5. Participant has a history of hypersensitivity to any component of the study intervention.
6. Participant had another primary malignancy within the previous 3 years.
7. Participants who require systemic steroid therapy 10 mg/day prednisone or another steroid equivalent dose.
8. Participants who have had a history of allogeneic organ transplant or any form of cell therapy involving prior conditioning chemotherapy within the past 20 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2032-06 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Up to 30 days
  The frequency and severity of treatment emergent adverse events and serious adverse events will be assessed when IOV-3001 administered
Recommended Dose for Phase 2 | Up to 30 days
  Determine the recommended dose for Phase 2

SECONDARY OUTCOMES:
Pharmacokinetics (PK) profile of IOV-3001 | Up to 8 days
  PK as measured by maximum observed drug concentration in plasma (Cmax) after single dose, and area under the concentration vs. time curve (AUC) after single dose.
Pharmacodynamic (PD) Profile of IOV-3001 | Up to 8 days
  The PD profile will be assessed by evaluating changes in the expression of phenotypic markers, serum cytokines and chemokines in blood.
Antidrug Antibody (ADA) Profile | Up to 5 years
  ADAs to IOV-3001 will be measured in blood.
Overall Response Rate (ORR) | Up to 5 years
  ORR is defined as the proportion of participants who have a confirmed CR or PR per RECIST v1.1 as assessed by the investigator from the date of lifileucel infusion until disease progression, start of a new anticancer therapy, or death due to any cause cause, whichever occurs first (up to a maximum of 5 years after the lifileucel infusion)
Complete Response (CR) rate | Up to 5 years
  CR rate is defined as the proportion of participants who have a confirmed CR per RECIST v1.1 as assessed by the investigator from the date of lifileucel infusion until disease progression, start of a new anticancer therapy, or death due to any cause cause (up to a maximum of 5 years after the lifileucel infusion)
Duration of Response (DOR) | Up to 5 years
  DOR is measured from the time that criteria are met for CR or PR per RECIST v1.1 as assessed by the investigator disease progression or death due to any cause (up to a maximum of 5 years after the lifileucel infusion)
Disease Control Rate (DCR) | Up to 5 years
  DCR is measured by the percentage of participants with a best overall confirmed response of CR or PR at any time participants with SD ≥ 4 weeks per RECIST v1.1 as assessed by the investigator from the date of lifileucel infusion disease progression, start of a new anticancer therapy, or death due to any cause (up to a maximum of 5 years after the lifileucel infusion)
Progression-Free Survival (PFS) | Up to 5 years
  PFS is defined as the time from the date of lifileucel infusion until disease progression per RECIST v1.1 as assessed by investigator or death due to any cause (up to a maximum of 5 years after the lifileucel infusion)
Overall Survival (OS) | Up to 5 years
  OS is the time from the date of lifileucel infusion to death due to any cause (up to a maximum of 5 years after the lifileucel infusion)
In vivo persistence of Lifileucel | Up to 5 years
  In vivo persistence of lifileucel products will be assessed in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Iovance Biotherapeutics Study Team, Study Director — Iovance Biotherapeutics
Locations (4):
- United States (3):
  - SCRI Oncology Partners- Denver, Denver, Colorado
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Greenslopes Private Hospital, Greenslopes, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No